CLINICAL TRIAL: NCT05087459
Title: Efficacy and Safety of Avatrombopag in Thrombocytopenia in Patients With Primary Hepatocellular Carcinoma Undergoing Elective Hepatectomy: a Multicenter, Randomized, Controlled Study
Brief Title: Treatment of Avatrombopag for Thrombocytopenia in Patients Undergoing Selective Resection of Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SKX-2005
Record Dates: First submitted 2021-09-28; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Thrombocytopenia
Keywords: Avatrombopag; Primary hepatocellular carcinoma; elective hepatectomy
MeSH Terms: conditions — Thrombocytopenia; Carcinoma, Hepatocellular | interventions — avatrombopag

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with primary hepatocellular carcinoma undergoing elective hepatectomy: The baseline platelet count before enrollment was < 75×10^9/L and > 30×10^9/L.The primary clinical diagnosis of hepatocellular carcinoma was confirmed, and the CNLC stages were Ia and Ib.An elective hepatectomy, including laparotomy or laparoscopic hepatectomy, except hepatectomy combined with splenectomy or radiofrequency ablation.
  Interventions: Drug: Avatrombopag

INTERVENTIONS:
Drug: Avatrombopag — On the basis of conventional treatment, Avatrombopag was added, 30×10^9/L < platelet count < 50×10^9/L patients received Avatrombopag 60mg/d, 50×10^9/L≤ platelet count < 75×10^9/L patients received Avatrombopag 40mg/d for 5 consecutive days, and waited for a period of time after drug withdrawal.Surgery is expected to take place on day 10-13 of the initial dose.
  Other Names: Doptelet

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the most common malignant tumors in the world, accounting for the second leading cause of cancer death in China.Surgical treatment of hepatocellular carcinoma is the most important means for long-term survival of patients with hepatocellular carcinoma, including hepatectomy and liver transplantation.Chronic liver disease caused by hepatitis B infection is the main pathogenic factor of liver cancer in China. Meanwhile, nearly 80% of patients with hepatocellular carcinoma are complicated with cirrhosis, and the incidence of thrombocytopenia in patients with cirrhosis is reported to be as high as 78%.Many previous studies have found that thrombocytopenia is closely related to perioperative outcome of hepatocellular carcinoma.The purpose of this study was to evaluate the efficacy and safety of avatripopa in the treatment of thrombocytopenia in patients with primary hepatocellular carcinoma undergoing elective hepatectomy and its effect on perioperative outcome.

DETAILED DESCRIPTION:
The indicators included changes in platelet count before and after drug treatment and operation, the nature and amount of postoperative drainage (ascites), duration of indwelling drainage tube, intraoperative blood loss, perioperative complications, length of hospital stay, etc.After comprehensive consideration of all perioperative indicators, we selected the total amount of drainage (ascites) multiple days after surgery as the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand this study and be willing to abide by all research procedures and sign informed consent voluntarily before screening;
2. Male or female, at least 18 years old when signing informed consent;
3. The initial clinical diagnosis of hepatocellular carcinoma was confirmed, and the CNLC stages were IA and IB;
4. Before enrollment, baseline platelet count < 75×10^9/L and > 30×10^9/L;
5. Elective hepatectomy is proposed, including laparotomy or laparoscopic hepatectomy, except hepatectomy combined with splenectomy or radiofrequency ablation;
6. Child-pugh GRADE A;
7. HBsAg and/or anti-HCV positive;
8. Male patients who are infertile or who agree to use appropriate contraceptive methods from the beginning of screening until the completion of the post-treatment phase;
9. Women who have not undergone menopause or surgical sterilization need to agree to use highly effective contraception from the beginning of screening until the completion of the post-treatment phase;
10. According to the opinions of researchers, those who can meet the requirements of this study.

Exclusion Criteria:

1. Any diseases below: Solid malignancies other than hepatocellular carcinoma, blood system tumor, aplastic anemia, myelodysplastic syndrome, myelofibrosis, congenital thrombocytopenia, drug-induced thrombocytopenia, immune thrombocytopenia, need treatment of systemic infection (except viral hepatitis);
2. Always thrombosis or current or former state (such as cerebral infarction, myocardial infarction, angina pectoris, coronary artery carotid stenting and angioplasty, coronary artery bypass grafting, congestive heart failure, known to increase the risk of thromboembolic events of arrhythmias such as atrial fibrillation, pulmonary thromboembolism, deep vein thrombosis or diffuse intravascular coagulation syndrome).
3. A known history of hereditary prethrombotic syndrome (e.g., clotting factor V Leiden mutation, prothrombin G20210A mutation, or hereditary antithrombin III (ATIII) deficiency);
4. Transfusion of platelets or blood products containing platelets within 7 days prior to screening;
5. Use erythropoietin within 7 days before screening;
6. Rhil-11,rhTPO, TPO receptor agonists (such as Avatriprap, altrippal, or romistetine) or splenic embolization within 30 days prior to screening;
7. Use of any of the following drugs or treatments within 90 days prior to screening: chemotherapy, interferon preparations, radiation;
8. Patients requiring systemic chemotherapy, targeted therapy, immunotherapy, traditional Chinese herbal therapy or radiation therapy during the study period;
9. At screening time, hemoglobin level ≤9.0g/dL or ≥18.0g/dL in male patients and > 15.0g/dL in female patients, and hematocrit in male ≥0.54 and female ≥0.45;
10. Bleeding score ≥2 at screening (according to the WHO Bleeding scale);
11. Pt-inr and APTT at screening were lower than 80% of the lower limit of normal range or higher than 120% of the upper limit of normal range;
12. Preoperative anticoagulant or antiplatelet therapy should not be suspended according to the standard (low-dose aspirin is allowed to continue);
13. Female subjects who are breast-feeding or pregnant at the time of screening, or who plan to become pregnant during the study period;
14. Known or suspected persistent alcohol or drug abuse;
15. Known allergy to Avatripopa or any of its excipients;
16. HIV infected persons;
17. Participate in another clinical study within 30 days prior to screening, using any exploratory drugs or devices;Allowed to participate in observational studies;
18. The investigator believes that the accompanying medical history may affect the subjects' safe completion of the study;
19. In the opinion of the investigator, there are any other factors that may not be suitable for inclusion or affect participation or completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective hepatectomy with thrombocytopenia in adults with primary hepatocellular carcinoma
Sampling Method: Probability Sample
Enrollment: 141 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with a platelet count ≥75×10^9/L and an increase of platelet count more than 20% from baseline | on day 9-12 of treatment
  The Percentage of patients in the treatment group with platelet count ≥75×10^9/L (the highest test value of of platelet count was taken on day 9-12 of treatment) and an increase of platelet count more than 20% from baseline before operation.
Comparison of total amount of postoperative drainage fluid between treatment group and control group | on day 1-5 after surgery
  Comparison of total amount of postoperative drainage fluid on day 1, 3 and 5 after surgery between treatment group and control group

SECONDARY OUTCOMES:
Comparison of intraoperative blood loss | During surgery
  Comparison of intraoperative blood loss between Treatment group and control group.
Proportion of patients receiving remedial treatment due to bleeding risk after surgery | on day 0-30 after surgery
  Comparison of the proportion of patients receiving remedial treatment due to bleeding risk after surgery between the treatment group and the control group
Indwelling time of drainage tube | on day 0-10 after surgery
  Comparison of postoperative indwelling time of drainage tube between treatment group and control group
Red blood cell count and hemoglobin content of drainage fluid | on day 1-5 after surgery
  Comparison of red blood cell count and hemoglobin content of drainage fluid between treatment group and control group on the 1st, 3rd and 5th day after operation
Postoperative hospitalization time | on 0-30 day after surgery
  Comparison of postoperative hospitalization time between treatment group and control group
Preoperative platelet count increase from baseline | before surgery
  Preoperative platelet count increase from baseline in treatment group.
The change of platelet count from baseline at different time points | through study completion, an average of 1 year
  The change of platelet count from baseline at different time points in the treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, MD PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller JB, Figueroa EJ, Haug RM, Shah NL. Thrombocytopenia in Chronic Liver Disease and the Role of Thrombopoietin Agonists. Gastroenterol Hepatol (N Y). 2019 Jun;15(6):326-332. PMID 31391802
- [Background] Li J, Han B, Li H, Deng H, Mendez-Sanchez N, Guo X, Qi X. Association of coagulopathy with the risk of bleeding after invasive procedures in liver cirrhosis. Saudi J Gastroenterol. 2018 Jul-Aug;24(4):220-227. doi: 10.4103/sjg.SJG_486_17. PMID 29956689